CLINICAL TRIAL: NCT03954600
Title: A Phase 1, Randomized, Double-Blind, Single and Multiple Ascending Dose Trial of the Safety, Tolerability and Pharmacokinetics of NPT520-34 in Healthy Subjects
Brief Title: A Study to Assess the Safety, Tolerability and PK of NPT520-34 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neuropore Therapies Inc. (Industry)
Collaborators: Celerion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NPT520-34-001
Record Dates: First submitted 2019-05-08; First posted 2019-05-17 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2019-05

CONDITIONS: Healthy Volunteers
Keywords: Phase 1; Safety; Tolerability; Pharmacokinetics; Parkinson's Disease; Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Parkinson Disease; Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- NPT520-34 - SAD Cohort 1, Dose 1 (Unfed) (Other): Single ascending dose of orally administered capsule(s) NPT520-34: 125 mg OR Single dose of orally administered placebo capsule(s) to match dose. Unfed.
  Interventions: Drug: NPT520-34 (125 mg); Drug: Placebos (125 mg)
- NPT520-34 - SAD Cohort 1, Dose 1 (Fed) (Other): Single ascending dose of orally administered capsule(s) NPT520-34: 125 mg OR Single dose of orally administered placebo capsule(s) to match dose. Fed.
  Interventions: Drug: NPT520-34 (125 mg); Drug: Placebos (125 mg)
- NPT520-34 - SAD Cohort 2, Dose 2 (Other): Single ascending dose of orally administered capsule(s) NPT520-34: 250 mg OR Single dose of orally administered placebo capsule(s) to match dose.
  Interventions: Drug: NPT520-34 (125 mg); Drug: Placebos (125 mg)
- NPT520-34 - SAD Cohort 3, Dose 3 (Other): Single ascending dose of orally administered capsule(s) NPT520-34: 500 mg OR Single dose of orally administered placebo capsule(s) to match dose.
  Interventions: Drug: NPT520-34 (125 mg); Drug: Placebos (125 mg)
- NPT520-34 - SAD Cohort 4, Dose 4 (Other): Single ascending dose of orally administered capsule(s) NPT520-34: 1000 mg OR Single dose of orally administered placebo capsule(s) to match dose.
  Interventions: Drug: NPT520-34 (125 mg); Drug: Placebos (125 mg)
- NPT520-34 - MAD Cohort 1, Dose 1 (Other): Multiple ascending dose of orally administered capsule(s) NPT520-34: TBD mg OR Single dose of orally administered placebo capsule(s) to match dose.
  Interventions: Drug: NPT520-34 (125 mg); Drug: Placebos (125 mg)
- NPT520-34 - MAD Cohort 2, Dose 2 (Other): Multiple ascending dose of orally administered capsule(s) NPT520-34: TBD mg OR Single dose of orally administered placebo capsule(s) to match dose.
  Interventions: Drug: NPT520-34 (125 mg); Drug: Placebos (125 mg)
- NPT520-34 - MAD Cohort 3, Dose 3 (Other): Multiple ascending dose of orally administered capsule(s) NPT520-34: TBD mg OR Single dose of orally administered placebo capsule(s) to match dose.
  Interventions: Drug: NPT520-34 (125 mg); Drug: Placebos (125 mg)

INTERVENTIONS:
Drug: NPT520-34 (125 mg) — NPT520-34, 125 mg oral capsules (size 1)
Drug: Placebos (125 mg) — Placebo, 125 mg oral capsules

SUMMARY:
To evaluate the PK, safety and tolerability of orally administered NPT520-34 in healthy subjects at single and multiple doses that may be therapeutically relevant.

ELIGIBILITY:
Inclusion Criteria:

1. informed of, and willing and able to comply with, all of the protocol requirements and the investigational nature of the study, and have signed an informed consent form in accordance with institutional and regulatory guidelines;
2. male or female adults between 18 and 55 years of age, inclusive;
3. female subjects must be of non-childbearing potential (i.e. post-menopausal for at least 2 years) or surgically sterile (hysterectomy, bilateral oophorectomy, tubal ligation) or nonsurgically sterile (hysteroscopic sterilization, i.e. Essure);
4. male subjects must be willing to use an adequate barrier method of contraception for the duration of the study and for 90 days after dosing and no sperm donations for the duration of the study and for 90 days after dosing. Male subjects who are surgically sterile (16 weeks post-surgery, or documented proof of Post-Vasectomy Semen Analysis (PVSA) with negative sperm results) need not employ a method of contraception;
5. non-smokers for at least six months;
6. BMI = 18.0 - 32.0 kg/m2 inclusive;
7. in good health, in the judgment of the Investigator, as determined by: 7a. medical history indicative of no serious or severe chronic conditions requiring frequent medical intervention or continual pharmacologic management, and no medical or social conditions that would potentially interfere with the subject's ability to comply with the study visit schedule or the study assessments; 7b. no clinically significant abnormalities in body temperature, heart rate, respiratory rate, blood pressure; 7c. no clinically significant abnormalities in the 12-lead electrocardiogram (ECG); 7d. no clinically significant abnormalities in clinical chemistry (ALT, AST, total bilirubin must be at or below the upper limit of normal and eGFR must be ≥ 90 mL/min), hematology (hemoglobin ≥ 11.5 g/dL for females and ≥ 13 g/dL for males), coagulation and urinalysis; lab tests may be repeated, if necessary (details are provided in the attached flow chart of study assessments).
8. negative results on the following screening laboratory tests: urine drug screen, urine alcohol screen, serum pregnancy test, hepatitis B surface antigen, hepatitis C antibody, and human immunodeficiency virus antibody.

Exclusion Criteria:

1. females of child bearing potential
2. history of a significant medical condition, including cholecystectomy or clinically significant GI tract resection, that may interfere with absorption, distribution or elimination of NPT520-34, or with the clinical and laboratory safety assessments in this study;
3. history of pre-existing thyroid abnormalities, such as hyper or hypothyroidism;
4. history of lactose intolerance;
5. history of drug hypersensitivity and disorders affecting respiratory function (e.g., COPD, asthma) and cardiac disorders predisposing to cardiac adverse events
6. history of or current alcohol abuse and/or other drug addiction < 2 years prior to screening, or a positive urine drug or alcohol screen (e.g., amphetamines, barbiturates, benzodiazepines, opiates, cannabinoids, alcohol and cocaine);
7. positive for HBVsAg, HCV Ab, HIV Ab;
8. 12 lead ECG showing the following: having a corrected QTc interval > 450 msec or <340 msec (Fridericia's correction);
9. sustained supine systolic blood pressure > 140 or < 90 mm Hg or supine diastolic blood pressure > 90 or < 50 mm Hg at Screening or Day -1. The average of the 2 assessments of BP taken at each visit will be used to exclude a subject;
10. resting pulse rate at screening of > 100 or < 45.
11. donated or lost > 500 mL of blood < 56 days prior to enrollment into this study;
12. plasma donation within 7 days prior to enrollment into this study;
13. active infection or febrile illness < 14 days prior to the first dose of study medication;
14. use of prescription (including hormone replacement therapy) or over-the-counter medications or herbal supplements ≤ 14 days prior to dosing and until completion of follow-up visit on Day 7 for the SAD subjects and Day 21 for the MAD subjects;
15. excessive regular caffeine intake (>250 mg of caffeine per day);
16. have participated in other clinical studies of a new chemical entity within 30 days prior to admission to the CRU.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2019-05-05 (Actual); Primary Completion 2019-10-02 (Actual); Study Completion 2019-10-09 (Actual)

PRIMARY OUTCOMES:
Safety/Tolerability of Single Ascending Doses (125 mg, 250 mg, 500 mg and 1000 mg) | Baseline, Day 1, 2 3, 5 and 7
  A) Incidence of clinically significant treatment-emergent changes in the following clinical measures: 1) physical examination, 2) suicidal ideation, 3) vital signs 4) continuous telemetry for 1 hour prior to dosing and for 2 hours post-dose, 5) continuous telemetry for 1 hour prior to dosing and for 2 hours post-dose.
  B) Incidence in clinical significant treatment-emergent changes in the following laboratory measures: 1) hematology, 2) clinical chemistry, 3) FSH (post-menopausal women only), 4) coagulation, 5) urinalysis
  C) Incidence of treatment-emergent adverse events
  D) Incidence of treatment-emergent serious adverse events
Maximum observed plasma concentration of Single Ascending Doses (125 mg, 250 mg, 500 mg and 1000 mg) | Day 1, 2, 3, 5, 7
  Noncompartmental calculation of maximum observed plasma concentration (Cmax);
Time to maximum plasma concentration of Single Ascending Doses (125 mg, 250 mg, 500 mg and 1000 mg) | Day 1, 2, 3, 5, 7
  Noncompartmental calculation of time to maximum plasma concentration (Tmax);
Area under the plasma concentration-time curve from 0 hour to the time of the last quantifiable plasma concentration of Single Ascending Doses (125 mg, 250 mg, 500 mg and 1000 mg) | Day 1, 2, 3, 5, 7
  Noncompartmental calculation of area under the plasma concentration-time curve from 0 hour to the time of the last quantifiable plasma concentration [AUCt];
Area under the plasma concentration-time curve extrapolated to infinity of Single Ascending Doses (125 mg, 250 mg, 500 mg and 1000 mg) | Day 1, 2, 3, 5, 7
  Noncompartmental calculation of area under the plasma concentration-time curve extrapolated to infinity (AUCinf) after dosing
Apparent oral clearance of Single Ascending Doses (125 mg, 250 mg, 500 mg and 1000 mg) | Day 1, 2, 3, 5, 7
  Noncompartmental calculation of apparent oral clearance (CL/F)
Apparent oral volume of distribution during the terminal phase of Single Ascending Doses (125 mg, 250 mg, 500 mg and 1000 mg) | Day 1, 2, 3, 5, 7
  Noncompartmental calculation of apparent oral volume of distribution during the terminal phase (Vz/F)
Mean residence time of Single Ascending Doses (125 mg, 250 mg, 500 mg and 1000 mg) | Day 1, 2, 3, 5, 7
  Noncompartmental calculation of mean residence time (MRT)
Terminal elimination half-life of Single Ascending Doses (125 mg, 250 mg, 500 mg and 1000 mg) | Day 1, 2, 3, 5, 7
  Noncompartmental calculation of terminal elimination half-life (T½);
Safety/Tolerability as measures of hematology, clinical chemistry, FSH, coagulation and urinalysis of multiple ascending doses (250 mg and 500 mg) | Baseline, Day 2, 4, 7, 11, 12, 13, 14, and 21
  A) Incidence in clinical significant treatment-emergent changes in hematology
  B) Incidence in clinical significant treatment-emergent changes in clinical chemistry
  C) Incidence in clinical significant treatment-emergent changes in FSH (post-menopausal women only)
  D) Incidence in clinical significant treatment-emergent changes in coagulation
  E) Incidence in clinical significant treatment-emergent changes in urinalysis
Safety/Tolerability as measures of vital signs and physical examination of multiple ascending doses (250 mg and 500 mg) | Baseline, Day 1, 2, 7, 8, 9, 10, 11, 14, 16, 18 Day 21
  A) Incidence of clinically significant treatment-emergent changes in vital signs
  B) Incidence of clinically significant treatment-emergent changes in physical examination
Safety/Tolerability as measures of continuous telemetry of multiple ascending doses (250 mg and 500 mg) | Baseline, Day 1, 2, 7, 8, 9, 10, 11, 14, and 15
  A) Incidence of clinically significant treatment-emergent changes in continuous telemetry
Safety/Tolerability as measures of suicidal ideation, 12-lead ECG, adverse events and serious adverse events of multiple ascending doses (250 mg and 500 mg) | Baseline, Day 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 16, 18 Day 21
  A) Incidence in clinical significant treatment-emergent changes in suicidal ideation
  B) Incidence in clinical significant treatment-emergent changes in 12-lead ECG
  C) Incidence of treatment-emergent adverse events
  D) Incidence of treatment-emergent serious adverse events
Safety/Tolerability as measure of continuous ECG of Multiple Ascending Doses (250 mg and 500 mg) | Baseline, Day 1, 7, and 14
  A) Incidence in clinical significant treatment-emergent changes in continuous ECG telemetry
Maximum observed plasma concentration (Cmax) after dosing on Day 1 of Multiple Ascending Doses (250 mg, 500 mg) | Baseline, Day 1 and 2
  Noncompartmental calculation of maximum observed plasma concentration (Cmax) after dosing on Day 1
Maximum observed concentration at steady-state after dosing on Day 14 of Multiple Ascending Doses (250 mg, 500 mg) | Day 14
  Noncompartmental calculation of maximum observed concentration at steady-state after dosing on Day 14
Concentration observed at the end of the dosing interval of Multiple Ascending Doses (250 mg, 500 mg) | Day 14, 16, 18
  Noncompartmental calculation of concentration observed at the end of the dosing interval (Ctrough)
Time to max. plasma concentration after dosing on Day 1 of Multiple Ascending Doses (250 mg, 500 mg) | Day 1
  Noncompartmental calculation of time to max. plasma concentration after dosing on Day 1
Time to reach Cmax,ss of Multiple Ascending Doses (250 mg, 500 mg) | Day 14, 16, 18 and 21
  Noncompartmental calculation of time to reach Cmax,ss
Area under the plasma concentration-time curve from 0 hour to the time of the last quantifiable plasma concentration of Multiple Ascending Doses (250 mg, 500 mg) | Baseline, Day 1, 2, 7, 8, 9, 10, 11, 14, 16, 18 and 21
  Noncompartmental calculation of area under the plasma concentration-time curve from 0 hour to the time of the last quantifiable plasma concentration (AUCt)
Area under the plasma concentration-time curve extrapolated to infinity after dosing of Multiple Ascending Doses (250 mg, 500 mg) | Baseline, Day 1, 2, 7, 8, 9, 10, 11, 14, 16, 18 and 21
  Noncompartmental calculation of area under the plasma concentration-time curve extrapolated to infinity after dosing (AUCinf)
Area under the concentration time curve from 0-24 hours after dosing on Day 1 of Multiple Ascending Doses (250 mg, 500 mg) | Day 1
  Noncompartmental calculation of the area under the concentration time curve from 0-24 hours after dosing on Day 1 (AUC0-24)
The area under the concentration time curve during a dosing interval (tau) at steady state after dosing on Day 14 of Multiple Ascending Doses (250 mg, 500 mg) | Baseline, Day 1, 2, 7, 8, 9, 10, 11, 14, 16, 18 and 21
  Noncompartmental calculation of the area under the concentration time curve during a dosing interval (tau) at steady state after dosing on Day 14 (AUCtau)
Apparent oral clearance of Multiple Ascending Doses (250 mg, 500 mg) | Day 1
  Noncompartmental calculation of apparent oral clearance (CL/F)
Apparent total plasma clearance after oral administration, calculated as Dose/AUCtau after dosing on Day 14 of Multiple Ascending Doses (250 mg, 500 mg) | Day 14
  Noncompartmental calculation of apparent total plasma clearance after oral (extravascular) administration (CL,ss/F), calculated as Dose/AUCtau after dosing on Day 14
Apparent oral volume of distribution during the terminal phase of Multiple Ascending Doses (250 mg, 500 mg) | Day 14, 16, 18 and 21
  Noncompartmental calculation of apparent oral volume of distribution during the terminal phase (Vz/F)
Mean residence time of Multiple Ascending Doses (250 mg, 500 mg) | Baseline, Day 1, 2, 7, 8, 9, 10, 11, 14, 16, 18 and 21
  Noncompartmental calculation of mean residence time (MRT)
Terminal elimination half-life of Multiple Ascending Doses (250 mg, 500 mg) | Day 14, 16, 18 and 21
  Terminal elimination half-life

SECONDARY OUTCOMES:
Maximum Tolerated Dose of Single Ascending Doses (125 mg, 250 mg, 500 mg and 1000 mg) | Day 1, 2, 3, 5, Day 7
  A) 2/6 subjects assigned to NPT520-34 have SAEs or Grade ≥3 lab abnormalities, considered related to study drug B) 1/6 subjects assigned to NPT520-34 has liver function tests, which: 1) ALT or AST>3x ULN or bilirubin >1.5x ULN and related to study drug C) 1/6 subjects assigned to NPT520-34 have liver function tests, which: 1) ALT or AST>3x ULN or bilirubin>1.5x ULN and related to study drug D) 1/ 6 subjects assigned to NPT520-34 have kidney function tests, which: 1) eGFR<60 mL/min and relationship to study drug is considered related, 2) serum creatinine>2x above baseline and relationship to study drug is considered related E) 2/ 6 subjects assigned to NPT520-34 have kidney function tests, which: 1) eGFR<60 mL/min and related to study drug, 2) serum creatinine > 2x above baseline and related to study drug F) Any subject experiences a SAE related to study drug G) Further dose escalation poses inappropriate safety risk according to Sponsor/Investigator
Maximum Tolerated Dose of Multiple Ascending Doses (250 mg and 500 mg) | Baseline, Day 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 16, 18 Day 21
  A) 2/6 subjects assigned to NPT520-34 have SAEs or Grade ≥3 lab abnormalities, considered related to study drug B) 1/6 subjects assigned to NPT520-34 has liver function tests, which: 1) ALT or AST>3x ULN or bilirubin >1.5x ULN and related to study drug C) 1/6 subjects assigned to NPT520-34 have liver function tests, which: 1) ALT or AST>3x ULN or bilirubin>1.5x ULN and related to study drug D) 1/ 6 subjects assigned to NPT520-34 have kidney function tests, which: 1) eGFR<60 mL/min and relationship to study drug is considered related, 2) serum creatinine>2x above baseline and relationship to study drug is considered related E) 2/ 6 subjects assigned to NPT520-34 have kidney function tests, which: 1) eGFR<60 mL/min and related to study drug, 2) serum creatinine > 2x above baseline and related to study drug F) Any subject experiences a SAE related to study drug G) Further dose escalation poses inappropriate safety risk according to Sponsor/Investigator

OTHER OUTCOMES:
Exploratory Biomarkers of Single Ascending Doses (125 mg, 250 mg, 500 mg and 1000 mg) | Baseline, Day 1, 2, Day 7
  To assess the following exploratory biomarkers: DHEA-S, DHEA, Cortisol Free, Copeptin, Osmolality Serum, Prolactin, FSH, LH, TSH, T3 Free, T4 free, Prostaglandin E2, Angiotensin II, Renin.
Exploratory Biomarkers of Multiple Ascending Doses (250 mg and 500 mg) | Baseline, Day 1, Day 7, 14, and 21
  To assess the following exploratory biomarkers: DHEA-S, DHEA, Cortisol Free, Copeptin, Osmolality Serum, Prolactin, FSH, LH, TSH, T3 Free, T4 free, Prostaglandin E2, Angiotensin II, Renin.

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Armas, M.D., Principal Investigator — Celerion
Locations (1):
- Celerion, Inc, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No